CLINICAL TRIAL: NCT04172974
Title: Screening and Managing Depression and Anxiety with Therapist-assisted EHealth Intervention in Patients with Ischemic Heart Disease in the Cardiac Rehabilitation Setting
Brief Title: EHealth Intervention to Manage Depression and Anxiety in Patients with Ischemic Heart Disease
Acronym: eMindYourHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: OPEN - Odense Patient data Explorative Network, The University of Southern Denmark, Odense, Denmark (Unknown)
Responsible Party: Principal Investigator, Susanne Schmidt Pedersen, Professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18/39431
Record Dates: First submitted 2019-10-31; First posted 2019-11-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Comparison of depression/anxiety treatment versus usual care
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment for depression and anxiety (Experimental): Treatment
  Interventions: Other: eHealth intervention
- Usual care (Other): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: eHealth intervention — Modules developed for depression and anxiety based on cognitive behavioral therapy (CBT), acceptance and commitment therapy (ACT) and compassion-focused coping
  Arms: Treatment for depression and anxiety
Other: Usual Care — Treatment according to national clinical guideline (referral to GP)
  Arms: Usual care

SUMMARY:
This study evaluates the effectiveness and cost-effectiveness of a therapy-assisted internet-based intervention in patients with ischemic heart disease and co-morbid depression and anxiety referred for cardiac rehabilitation. Half of the patients will receive the intervention and the other half usual care. We hypothesize that the intervention will lead to a reduction in patients' symptoms of depression and anxiety and be cost-effective.

DETAILED DESCRIPTION:
The 12-week intervention will consist of 9 modules and 2 optional modules that will be delivered to patients in the active intervention via a platform or app. Psychologists will provide asynchronous guidance via the platform. Motivational interviewing will be used during the intervention to prevent dropout. The psychologist may contact patients via telephone during the intervention if needed. All patients will have access to the intervention up to 6 months' post intervention so that they can revisit the material and reuse it on a need-to-basis. Patients will be recommended to use this option and to note specific time points in their agenda where they will access the intervention. A brief purpose-designed interview protocol that includes elements from the SCAN interview will be carried out by psychologists trained in conducting the interview.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of ischemic heart disease (diagnostic codes I20-I25)
* Referred for CR
* HADS score ≥ 8 on depression and or anxiety
* Access to a computer or smart phone
* Ability to use computer or smart phone
* Proficient in the Danish language
* Signing an informed consent form

Exclusion Criteria:

* Severe psychiatric disorder (i.e., borderline disorder, schizophrenia or bipolar disorder)
* Severe cognitive difficulties (e.g. severe brain damage, mental retardation, or dementia) that will prevent patients from participating
* Endorsement of suicidal ideation with daily suicidal thoughts (PHQ-9 item 9 >2)
* Participation in other intervention studies (unless they are clinical studies)
* Seeing a psychologist or mental health professional for the treatment of anxiety and depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Symptoms of depression | 3 months
  Measured by Hospital Anxiety and Depression Scale (range 0-21 - high score = more symptoms)

SECONDARY OUTCOMES:
Symptoms of anxiety | 3 months
  Measured by Hospital Anxiety and Depression Scale (range 0-21 - high score = more symptoms)
Symptoms of depression | 6 months
  Measured by Hospital Anxiety and Depression Scale (range 0-21 - high score = more symptoms)
Symptoms of anxiety | 6 months
  Measured by Hospital Anxiety and Depression Scale (range 0-21 - high score = more symptoms)
Symptoms of depression | 12 months
  Measured by Hospital Anxiety and Depression Scale (range 0-21 - high score = more symptoms)
Symptoms of anxiety | 12 months
  Measured by Hospital Anxiety and Depression Scale (range 0-21 - high score = more symptoms)
Patient-reported quality of life | 3 months
  Measured by the Health-related quality of life questionnaire (HeartQoL) - The measure consists of a global, physical and emotional sub scale. Score range is from 0-3 (high score = better QoL)
Patient-reported quality of life | 6 months
  Measured by the Health-related quality of life questionnaire (HeartQoL) - The measure consists of a global, physical and emotional sub scale. Score range is from 0-3 (high score = better QoL)
Patient-reported Quality of life | 12 months
  Measured by the Health-related quality of life questionnaire (HeartQoL) - The measure consists of a global, physical and emotional sub scale. Score range is from 0-3 (high score = better QoL)
Dropout | 3 months
  Number of patients dropped out in each arm
Cost-effectiveness | 3 months
  EUROQOL - 5 Questions with 5 levels with level 5 being the worst level
Cost-effectiveness | 6 months
  EUROQOL - 5 Questions with 5 levels with level 5 being the worst level
Cost-effectiveness | 12 months
  EUROQOL - 5 Questions with 5 levels with level 5 being the worst level
Perceived Stress | 3 months
  Measured with the Perceived Stress Scale (range 0-40 - high score = highest level of stress)
Perceived Stress | 6 months
  Measured with the Perceived Stress Scale (range 0-40 - high score = highest level of stress)
Perceived Stress | 12 months
  Measured with the Perceived Stress Scale (range 0-40 - high score = highest level of stress)
Health complaints | 3 months
  Measured with the Health Complaints Scale (range 0-95 - 95=worse health)
Health complaints | 6 months
  Measured with the Health Complaints Scale (range 0-95 - 95=worse health)
Health complaints | 12 months
  Measured with the Health Complaints Scale (range 0-95 - 95=worse health)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne S Pedersen, PhD, Principal Investigator — University of Southern Denmark
Locations (13):
- Denmark (13):
  - Aalborg University Hospital, Aalborg
  - Helle Lynge Kanstrup, Aarhus
  - Herlev / Gentofte Hospital, Herlev
  - Regionshospital Nordjylland, Hjørring
  - Holbæk Hospital, Holbæk
  - Holbæk Sygehus, Holbæk
  - Sygehus Lillebælt Kolding, Kolding
  - Odense University Hospital (Odense), Odense
  - Randers Municipality, Randers
  - Zealand University Hospital, Roskilde
  - Odense University Hospital (Svendborg), Svendborg
  - Sygehus Lillebælt, Vejle
  - Vordingborg Municipality, Vordingborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen SS, Andersen CM, Ahm R, Skovbakke SJ, Kok R, Helmark C, Wiil UK, Schmidt T, Olsen KR, Hjelmborg J, Zwisler AD, Frostholm L. Efficacy and cost-effectiveness of a therapist-assisted web-based intervention for depression and anxiety in patients with ischemic heart disease attending cardiac rehabilitation [eMindYourHeart trial]: a randomised controlled trial protocol. BMC Cardiovasc Disord. 2021 Jan 7;21(1):20. doi: 10.1186/s12872-020-01801-w. PMID 33413109